CLINICAL TRIAL: NCT02414984
Title: Registry of Patients With Rheumatoid Arthritis Exposed to Golimumab (Go-Compl-Ar): Review and Analysis of Compliance in Colombia
Brief Title: Registry for Analysis of Compliance in Colombian Participants With Rheumatoid Arthritis Exposed to Golimumab
Acronym: Go-Compl-Ar
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment (Terminated due to lack of patient recruitment)
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR105492; CNTO148ARA4004 (Other: Janssen-Cilag, S.A.)
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Golimumab; Observational; Compliance
MeSH Terms: conditions — Arthritis, Rheumatoid; Patient Compliance | interventions — golimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Golimumab: Participants with rheumatoid arthritis in Colombia, for whom the treating physician has decided to treat with golimumab prior to enrolment. All participants will be observed for 24 months. Any changes including addition of new medications or dose modifications of existing medications will be entirely according to the treating physician's judgment.
  Interventions: Biological: Golimumab

INTERVENTIONS:
Biological: Golimumab — This is an observational study. Participants with rheumatoid arthritis in Colombia will be observed for 24 months.
  Other Names: CNTO148

SUMMARY:
The purpose of this study is to describe adherence to golimumab in Colombian participants with rheumatoid arthritis (RA) experiencing adequate treatment response, in a real-world clinical settings.

DETAILED DESCRIPTION:
This is a multi-center (when more than one hospital or medical school team work on a medical research study), non-interventional, prospective cohort study that will enroll participants with RA in Colombia, for whom the treating physician has decided to treat with golimumab prior to enrolment. All participants will be observed for adherence to golimumab treatment for 24 months from study start (Week 0), and recommended follow up assessments will be every 3 months. Any changes including addition of new medications or dose modifications of existing medications will be entirely according to the treating physician's judgment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe RA for whom the physician had decided to treat with golimumab according to the local product label, with the first dose being administered between 12 and 26 weeks prior to study enrollment
* Participants who have achieved an adequate therapeutic response to regular doses of golimumab, within 12 to 26 weeks of treatment
* Participants should be evaluated for tuberculosis (TB) exposure/risk factors or managed for active and latent TB (per local requirements and according to the local product label)
* Participants who have been evaluated for active/latent hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Participants for whom, since golimumab initiation, a complete medical record is available

Exclusion criteria:

* Participants who have received and terminated golimumab treatment in the past
* Participants that have been treated with golimumab for more than 26 weeks prior to enrolment in the study
* Participants with use of any other investigational agent less than or equal to 30 days before starting treatment with golimumab
* Participants with suspected latent TB, having not received prophylactic treatment of at least 4 weeks
* Participants with suspected or active TB
* Participants with active/latent HBV or HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of Colombian rheumatoid arthritis participants, who have been prescribed golimumab by their treating physician prior to, and independently of, study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Treatment Adherence Measured by Continuous Measures of Medication Gaps (CMG) | 24 months
  Adherence rates to golimumab will be measured by the Continuous Measures of Medication Gaps (CMG). CMG provides an approximate percentage of time in which a participant is without medication available for use. Number of days of delay between consecutive golimumab injections will be observed throughout the study.

SECONDARY OUTCOMES:
Frequency of Treatment Suspension | 24 months
  Treatment suspension is defined as a treatment gap of at least 2 cycles of golimumab, with subsequent restart, as assessed by CMG.
Number of Treatment Termination | 24 months
  Treatment termination is defined as a treatment gap of at least 2 cycles of golimumab, with no treatment restart as assessed by CMG.
Change From Baseline in 28-Joint Disease Activity Score (DAS-28) at Month 6, 12, 18, and 24 or Early Termination | Baseline, Month 6, 12, 18, and 24 or Early Termination
  DAS28 is calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) or the C-reactive protein (CRP) and patient's global assessment (PtGA) of disease activity (participant rate arthritis activity using visual analog scale [VAS] ranging from 0 to 100; higher scores indicated greater affectation due to disease activity).
Change From Baseline in Patient's Global Assessment (PtGA) at Month 6, 12, 18, and 24 or Early Termination | Baseline, Month 6, 12, 18, and 24 or Early Termination
  Participant will rate arthritis activity using Visual Analog Scale (VAS) ranging from 0 to 100; higher scores indicated greater affectation due to disease activity.
Change From Baseline in Physician Global Assessment of Disease Activity (MDGA) at Month 6, 12, 18, and 24 or Early Termination | Baseline, Month 6, 12, 18, and 24 or Early Termination
  Physician will rate arthritis activity using Visual Analog Scale (VAS) ranging from 0 to 100; higher scores indicated greater affectation due to disease activity.
Change From Baseline in Work Related Productivity at Month 6, 12, 18, and 24 or Early Termination | Baseline, Month 6, 12, 18, and 24 or Early Termination
  Work related productivity (absenteeism, presenteeism, and impairment in daily activities) will be assessed using Work Productivity and Activity Impairment Questionnaire: Rheumatoid Arthritis (WPAI-RA), which consisted of 6 items: 1) Current employment status; 2) Number of hours missed due to a health problem; 3) Number of hours missed due to other reasons; 4) Hours actually worked; 5) Degree to which health affected productivity while working; 6) Degree to which health affected regular (non-work) activities.
Change From Baseline in Quality of Life at Month 12 and 24 or Early Termination | Baseline, Month 12 and 24 or Early Termination
  Quality of life will be assessed by 36-Item Short-Form Health Survey (SF-36). SF-36 is a generic quality of life questionnaire that assesses 8 health concepts: 1) Limitations in physical activities because of health problems; 2) Limitations in social activities because of physical or emotional problems; 3) Limitations in usual role activities because of physical health problems; 4) Bodily pain; 5) General mental health (psychological distress and well-being); 6) Limitations in usual role activities because of emotional problems; 7) Vitality (energy and fatigue); 8) General health perceptions.
Change From Baseline in Functional Status at Month 6, 12, 18, and 24 or Early Termination | Baseline, Month 6, 12, 18, and 24 or Early Termination
  Functional status will be assessed by Health Assessment Questionnaire-Disability Index (HAQ-DI). HAQ-DI is a self-administered questionnaire measuring the participant's functional ability. It consists of 20 items converging to 8 scales measuring daily living activities: dress/groom; arise; eat; walk; hygiene; reach; grip; and common daily activities over past week. The participant rate each activity as 0 = without any difficulty, 1 = some difficulty, 2 = much difficulty and 3 = unable. The final score ranges from 0 to 3 with higher scores indicating more disability.
Change from Baseline in Utilization of Health Care Resources at Month 3, 6, 9, 12, 15, 18, 21, and 24 or Early Termination | Baseline, Month 3, 6, 9, 12, 15, 18, 21, and 24 or Early Termination
  Utilization of Health Care Resources will be measured by the Consumption of Health Care Resources Questionnaire, which includes 8 questions related to the participant's use of health care resources related to RA: 1) Extra or unscheduled visits to the study doctor office/clinic, 2) Visits to another physician/healthcare professional (like nurse, therapist, physiotherapist), 3) Visits to hospital emergency room/ total duration of stay (hours), 4) Use of an ambulance service, 5) Admitted to a hospital/ total duration of stay (hours), 6) Visit to a specialist, 7) Complementary alternative therapy visits, 8) Out of pocket expenses related to RA (for example over-the-counter medication, payments for health care professionals, medical procedures or laboratory tests, medical devices, health care or extra help at home, transportation costs, differences in cost of prescription medication not covered by insurance).
Number of Participants with Adverse Events (AEs) Leading to Treatment Discontinuation | 24 months
Number of Participants with Serious adverse Events (SAE) | 24 months
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag, S.A. Clinical Trial, Study Director — Janssen-Cilag, S.A.
Locations (5):
- Colombia (5):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Cali
  - Medellín

IPD SHARING:
Plan to Share IPD: No